CLINICAL TRIAL: NCT04558424
Title: Randomized, Double -Blind, Placebo Controlled, Trial to Evaluate the Effect of Zinc and Ascorbic Acid Supplementation in COVID-19 Positive Hospitalized Patients in BSMMU
Brief Title: RCT,Double Blind, Placebo to Evaluate the Effect of Zinc and Ascorbic Acid Supplementation in COVID-19 Positive Hospitalized Patients in BSMMU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, elora sharmin, assistant professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BSMMU 2020
Record Dates: First submitted 2020-09-21; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — gluconic acid; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Criteria
  Inclusion Criteria:
  * ≥ 18 years presenting symptoms who test positive for COVID-19
  * Moderate to severe patients obtained consent
  * Hypoxic respiratory failure (saturation <90% on air at rest or increasing oxygen requirement)
  * Chest examination findings of bilateral crackles on auscultation or chest x-ray showing bilateral infiltrates
  * C-Reactive Protein > 50mg/L
  * women of childbearing potential who meet the above and have a negative pregnancy test.
  Exclusion Criteria:
  * Pregnant women: Current known pregnancy positive pregnancy test.
  * Lactating women.
  * Documented history of mental illnesses
  * Multi-organ failure
  * Severe ARDS (requiring ventilator support on presentation in the form of invasive or non-invasive ventilation)
  * Septic Shock
  * Drug allergy/intolerance
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Immediately after randomization, random numbers of the two sets will assigned as patients code number. One set will be designated as intervention group and another group will placebo group. Two sets of code number that belongs to the intervention group and placebo group will be written with patient's id number. this total procedure will be conducted by the person unrelated to this research. Thus, the participants, caregiver, outcome assessor and the analyst, who require being blind for such study will effectively blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will consist of 50 patients who will be treated with zinc and vitamin C at a dose of 220 mg and 1 gram orally daily for 10 days in addition to their standard treatment
  Interventions: Dietary Supplement: zinc gluconate and ascorbic acid
- Placebo group (Placebo Comparator): This group will consist of 50 patients who will receive placebo at a dose same dose for 10 days in addition to their standard treatment.
  Interventions: Dietary Supplement: zinc gluconate and ascorbic acid

INTERVENTIONS:
Dietary Supplement: zinc gluconate and ascorbic acid — This group will consist of 50 patients who will receive 220 mg zinc and 1gm ascorbic acid for 10 days in addition to their standard treatment.

SUMMARY:
The first COVID-19 case was identified on March 7, 2020. Since then, 4127 deaths of the total 3,40583 confirmed cases are reported in Bangladesh of August 26, 2020. this new virus there has been an increase in the number of pneumonia, which are characterized by fever, sore throat ,asthenia, dry cough, lymphopenia, prolonged prothrombin time, elevated lactic dehydrogenase and CRP and a tomographic imaging indicative of interstitial pneumonia (ground glass and patchy shadows). Severe disease occurs in 15% of the cases with COVID-19 and may progress to critical disease in only 5% of the cases with a high risk of mortality. Critical disease may present as acute respiratory failure secondary to Acute Respiratory Distress Syndrome mainstay of treatment is supportive. Recent studies have shown the efficacy of vitamin C and Zinc administration in patients hospitalized for sepsis in the setting of intensive wards in terms of mortality reduction. The use of vitamin C arises from the experimental evidence of its anti-inflammatory and antioxidant properties. Zinc is known to modulate antiviral and antibacterial immunity and regulate inflammatory response. Zn may possess protective effect as preventive and adjuvant therapy of COVID-19 through reducing inflammation, improvement of mucociliary clearance, prevention of ventilator induced lung injury, modulation of antiviral and antibacterial immunity. Severity assessment tools for identifying patients at risk of deterioration due to sepsis. The quick Sequential (Sepsis-related) Organ Failure Assessment tool is the recommended tool to screen patients with suspected infection outside the intensive care unit (one point for each of altered mentation, respiratory rate ≥22 and systolic blood pressure ≤100 mmHg, with a score ≥2 suggesting high risk for deterioration).More generic tools designed to predict deterioration regardless of etiology have also been designed, such as the National Early Warning Score , widely used in the English National Health Service, Access alertness, RR, blood pressure , heart rate, oxygen saturation and temperature with increasing values for more abnormal measurements. A score of ≥3 in any category or score ≥5 overall triggers urgent patient review.D isease specific tools, such as CURB65, are recommended by respiratory societies worldwide.Each of altered mentation, blood urea >7.0, RR ≥30, SBP <90 or diastolic BP ≤60 and age ≥65 scores one point, with scores ≥2 considered moderate- severe.

DETAILED DESCRIPTION:
In view of the emerging COVID-19 pandemic caused by SARS-coV-2 virus, the search for potential protective and therapeutic antiviral strategies is of particular and urgent interest. Despite the lack of clinical data, certain indications suggest that modulation of zinc status may be beneficial in COVID-19. The use of vitamin C could be effective in terms of mortality and outcomes in patients with covid-19 pneumonia. Zinc and vitamin C are the over the counter supplementation and other study shows the effect of this in respiratory tract infection. This type of study is not done in Bangladesh. So, this will give a baseline data for further study which will help the researcher.

C. Related with socio-economic development: Health economic analysis will be done by total duration of hospital stay in comparing with total cost during admission in hospital. Benefits of this analysis will consider the:

* Reduced the severity and symptoms which will decrease the risk of mortality among the patients.
* Duration of hospital stay will reduce the treatment cost and as well the price of this nutrients supplements is very low.
* Costs are measured by the recorded number of patients and duration of hospital stay in both study groups. Number and duration will be recorded.

  3. Work plan:

Methodology Types of study: Randomized double-blind placebo Controlled Trial Place of study: Department of pharmacology, Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka.

Study population:

Eligible participants for randomization are COVID-19 positive patients admitted in BSMMU

* Ages Eligible for Study: 18 Years and older (Adult, Older Adult)
* Sexes Eligible for Study: All
* Accepts Healthy Volunteers: No Criteria

Inclusion Criteria:

* ≥ 18 years presenting symptoms who test positive for COVID-19
* Moderate to severe patients obtained consent
* Hypoxic respiratory failure (saturation <90% on air at rest or increasing oxygen requirement)
* Chest examination findings of bilateral crackles on auscultation or chest x-ray showing bilateral infiltrates
* C-Reactive Protein > 50mg/L
* women of childbearing potential who meet the above and have a negative pregnancy test.

Exclusion Criteria:

* Pregnant women: Current known pregnancy positive pregnancy test.
* Lactating women.
* Documented history of mental illnesses
* Multi-organ failure
* Severe ARDS (requiring ventilator support on presentation in the form of invasive or non-invasive ventilation)
* Septic Shock
* Drug allergy/intolerance Sampling technique: Patients who meet the inclusion criteria and who provide consent will be randomized by online graph pad software by using computer.

Sample size:

Sample size calculation P1 (1-P1) + P2 (1-P2) × (Zα+ Zβ)2 N = (P1- P2)2 Where, N= sample size P1 = control group response 50 % P2= treatment group response 20% Zα = Z value at a definite level of significance1.96 at 5% level of significance Zβ = Z value at a definite power 1.28 at 90 % power (when β is 0.10)

0.5 (1-0.5) + 0.2 (1- 0.2) × (1.96+ 1.28)2 N= (0.5-0.2)2

= 48 According to this formula sample size will be 48 in each group. We estimate that the drop-out rate will be 5%, total 50 patients will be in each group

Study variables

1. Demographic variables:

* Age
* Sex
* Ethnicity
* Past medical history - Hypertension, use of ACEI or ARB, DM, IHD, COPD, CKD, Obesity (BMI) and Cancer
* Presenting symptoms (dry cough, productive cough, fever, sore throat, myalgia, lethargy, headache, breathlessness, nausea, diarrhea and any other)
* Baseline observations on day of initiating treatment (Day 0): oxygen saturation (SpO2), fraction of inspired oxygen (FiO2), SpO2/FiO2 ratio, respiratory rate, body temperature, neutrophil-lymphocyte ratio, C-Reactive Protein & findings of bilateral infiltrates on chest-x-ray.
* Follow-up observations after randomization on Day 1,2,3,4 and 5 for SpO2/FiO2 ratio, respiratory rate, body temperature and C-Reactive Protein
* Length of stay (in days)
* Use of ventilator support (invasive or non-invasive ventilation)
* Side effects of drugs
* In-patient mortality

Methods:

Each patient will give informed consent and demographic data (age, sex) will be obtained and documented. All patients will receive standard routine medical care throughout the study. After collecting baseline data patients will be assigned to respective group randomly. A compliance sheet will be maintained for each patient. Regularity of drug intake will be ensured and recorded in the patient's compliance sheets by research assistant. Patients will be asked to report for any adverse effects of the medication given during the period of study. The study will follow the principle of the declaration of Helsinki and of the world medical assembly. The study will be conducted after the approval of the protocol by the institutional review board (IRB). Each patient will be assured that the present therapy would not provide harm, however in case of any untoward effect, assurance would be provided for proper medical treatment and care from the part of the researcher. Each patient had complete right to withdraw from the study at any time during the research.

Recruitment procedure for patients according to symptoms and who consent to participate in the study will be randomly allocated immediately after hospital admission to one of two groups; intervention (I), or placebo group (P).

Pre-designed case record form (CRF) will be used for collecting data, which will also contain the result of the study. The information collected in the CRF will be reviewed and inconsistencies will be investigated and clarified. Data from case record forms will be anonymized and stored securely in a secure online web-based portal. The study outline is presented in Figure 1.

Study procedure:

Randomization - After determining the sample size, patients will randomly be allocated into two groups to the patient's enrollment for the study. Randomization will be done by online graph pad software by using computer. the software automatically generated two distinct sets of numbers after giving necessary inputs (sample size, sets of number). The online graph pad calculator equally distributed the patients into two comparable groups. The randomization will conduct by a competent third group person, a professor of this University who has no relationship with this study.

Blinding - Immediately after randomization, random numbers of the two sets will assigned as patients code number. One set will be designated as intervention group and another group will placebo group. Two sets of code number that belongs to the intervention group and placebo group will be written with patient's id number. this total procedure will be conducted by the person unrelated to this research. Thus, the participants, caregiver, outcome assessor and the analyst, who require being blind for such study will effectively blind.

Allocation cancelation: In order to prevent selection bias, concealment of allocation will be done. Third person allocated two distinct sets of random numbers into intervention group and placebo group. The allocation code written in two different paper document and preserved in two separate pen drive which will sealed within two different envelop. The sealed enveloped will be preserved to another two distinguished professors. So, intervention allocation will not be known to any person involve in the research.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years presenting symptoms who test positive for COVID-19
* Moderate to severe patients obtained consent
* Hypoxic respiratory failure (saturation <90% on air at rest or increasing oxygen requirement)
* Chest examination findings of bilateral crackles on auscultation or chest x-ray showing bilateral infiltrates
* C-Reactive Protein > 50mg/L
* women of childbearing potential who meet the above and have a negative pregnancy test.

Exclusion Criteria:

* Pregnant women: Current known pregnancy positive pregnancy test.
* Lactating women.
* Documented history of mental illnesses
* Multi-organ failure
* Severe ARDS (requiring ventilator support on presentation in the form of invasive or non-invasive ventilation)
* Septic Shock
* Drug allergy/intolerance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
symptoms reduction time frame | 28 days
  Number of days to reach a 50 percent reduction in the cumulative 0-36 symptom score with each symptom evaluated on a 0-3 scale. Assessed symptoms are Fever, Cough, Shortness of Breath, Fatigue, Muscle or body aches, Headache, New loss of taste, New loss of smell, Congestion or runny nose, Nausea, Vomiting, Diarrhea. Each patient will have a composite score ranging from 0-36/day

SECONDARY OUTCOMES:
Symptom Resolution: Fever | 28 days
  The number of days required to reach a score of 0 from the symptom category of fever based on a 0-3 scale: 0 = ≤98.6, 1 = >98.6- 100.6, 2 = > 100.6 - 102.6, 3 = >102.6
Symptom Resolution: Cough | 28 days
  The number of days required to reach a score of 0 from the symptom category of cough based on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe
Symptom Resolution: Fatigue | 28 days
  The number of days required to reach a score of 0 from the symptom category of shortness of breath based on a 0-3 scale: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities
Symptom Resolution: Muscle/body aches | 28 days
  The number of days required to reach a score of 0 from the symptom category of muscle/body aches based on a 0-3 scale: 1=mild muscle/body aches, 2=moderate muscle/body aches , 3=severe muscle/body aches.
Symptom Resolution: Headache | 28 days
  The number of days required to reach a score of 0 from the symptom category of headache based on a 0-3 scale: 1=mild headache, 2=moderate headache, 3=severe headache.
Symptom Resolution: New loss of taste | 28 days
  The number of days required to reach a score of 0 from the symptom category of new loss of taste based on a 0-3 scale: 1=mild loss of taste, 2=moderate loss of taste, 3=severe loss of taste.
Symptom Resolution: New loss of smell | 28 days
  The number of days required to reach a score of 0 from the symptom category of new loss of smell based on a 0-3 scale: 1=mild loss of smell, 2=moderate loss of smell, 3=severe loss of smell.
Symptom Resolution: Congestion/ runny nose | 28 days
  The number of days required to reach a score of 0 from the symptom category of congestion/runny nose on a 0-3 scale: 1=mild congestion/runny nose , 2=moderate congestion/runny nose , 3=severe congestion/runny nose .
Symptom Resolution: Nausea | 28 days
  The number of days required to reach a score of 0 from the symptom category of nausea on a 0-3 scale: 1=mild nausea, 2=moderate nausea, 3=severe nausea.
Symptom Resolution: Vomiting | 28 days
  The number of days required to reach a score of 0 from the symptom category of vomiting on a 0-3 scale: 1=mild vomiting, 2=moderate vomiting, 3=severe vomiting.
Symptom Resolution: Diarrhea | 28 days
  The number of days required to reach a score of 0 from the symptom category of diarrhea on a 0-3 scale: 1=mild diarrhea, 2=moderate diarrhea, 3=severe diarrhea.
Day 5 Symptoms | 28 days
  Total symptom composite score at day 5 of study supplementation: Symptom categories of fever based on a 0-3 scale: 0 = ≤98.6, 1 = >98.6- 100.6, 2 = > 100.6 - 102.6, 3 = >102; Cough on a 0-3 scale: 0 = no cough, 1 = mild, 2 = moderate, 3 = severe; Shortness of Breath on a 0-3: 0 = no shortness of breath, 1 = with moderate intensity exercise 2 = with walking on flat surface 3 = short of breath with getting dressed or daily activities; and Fatigue on a 0-3 scale: 0 = No fatigue/energetic, 1=mild fatigue, 2=moderate fatigue, 3=severe fatigue.
Severity of Symptoms | 28 days
  Differences in severity of symptoms between study arms
Adjunctive Medications | 28 days
  Differences in number of patients who were prescribed adjunctive medications for their diagnosis between study arms
Supplementation Side Effects | 28 days
  Differences in number of patients in study arms who experienced side effects from the supplements.

CONTACTS AND LOCATIONS:
Overall Officials: sharmin, Principal Investigator — bangabandhu sheikh mujib medical unuversity
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the journal authority and make public as part of the publication
Supporting Information: SAP, ICF, CSR
Time Frame: six month
Access Criteria: Available on public domain like figshare, researchgate and others